CLINICAL TRIAL: NCT01484197
Title: A Multi-centre, Randomized, Double-blind, Double-dummy, Multiple-dose, Crossover Study to Evaluate the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of Orally Inhaled Indacaterol Administered as Either PulmoSphere or Lactose-blend Powder Via the Concept1 Device in Adult Patients With Persistent Asthma
Brief Title: A Study to Evaluate the Effects of Indacaterol Maleate as a New Formulation in the Concept 1 Device
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CIDD001A2201; 2011-001825-25 (EudraCT Number)
Record Dates: First submitted 2011-11-15; First posted 2011-12-02 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
Keywords: Asthma; Indacaterol; QAB149
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 75 µg Indacaterol (LB) + Placebo (PoS) (Experimental): 75 µg indacaterol maleate lactose blend (LB) + placebo to indacterol PulmoSphereTM (PoS) delivered via the Concept1 device once daily in the morning for 7 days.
  Interventions: Drug: 75 µg indacaterol maleate (LB); Drug: placebo to indacaterol (PoS)
- 75 µg Indacaterol (PoS) + Placebo (LB) (Experimental): 75 µg indacaterol maleate PulmoSphereTM (PoS) + placebo to indacterol lactose blend (LB) delivered via the Concept1 device once daily in the morning for 7 days.
  Interventions: Drug: 75 µg indacaterol maleate (PoS); Drug: placebo to indacaterol (LB)
- 37.5 µg Indacaterol (PoS) + Placebo (LB) (Experimental): 37.5 µg indacaterol maleate PulmoSphereTM (PoS) + placebo to indacaterol lactose blend (LB) delivered via the Concept1 device once daily in the morning for 7 days.
  Interventions: Drug: 37.5 µg indacaterol maleate (PoS); Drug: placebo to indacaterol (LB)
- Placebo (LB) and Placebo (PoS) (Experimental): Placebo to indacaterol PulmoSphereTM (PoS) + placebo to indacaterol lactose blend (LB) delivered via the Concept1 device once daily in the morning for 7 days.
  Interventions: Drug: placebo to indacaterol (LB); Drug: placebo to indacaterol (PoS)

INTERVENTIONS:
Drug: 75 µg indacaterol maleate (LB) — 75 µg indacaterol maleate lactose blend (LB) delivered via the Concept1 device once daily in the morning for 7 days.
  Arms: 75 µg Indacaterol (LB) + Placebo (PoS)
Drug: 75 µg indacaterol maleate (PoS) — 75 µg indacaterol maleate PulmoSphereTM (PoS) delivered via the Concept1 device once daily in the morning for 7 days.
  Arms: 75 µg Indacaterol (PoS) + Placebo (LB)
Drug: 37.5 µg indacaterol maleate (PoS) — 37.5 µg indacaterol maleate PulmoSphereTM (PoS) delivered via the Concept1 device once daily in the morning for 7 days.
  Arms: 37.5 µg Indacaterol (PoS) + Placebo (LB)
Drug: placebo to indacaterol (LB) — Placebo to indacaterol lactose blend (LB) delivered via the Concept1 device once daily in the morning for 7 days.
  Arms: 37.5 µg Indacaterol (PoS) + Placebo (LB); 75 µg Indacaterol (PoS) + Placebo (LB); Placebo (LB) and Placebo (PoS)
Drug: placebo to indacaterol (PoS) — Placebo to indacaterol PulmoSphereTM (PoS) delivered via the Concept1 device once daily in the morning for 7 days.
  Arms: 75 µg Indacaterol (LB) + Placebo (PoS); Placebo (LB) and Placebo (PoS)

SUMMARY:
This study will assess the pharmacodynamics, safety, tolerability and pharmacokinetics of two different formulations of indacaterol maleate, both administered via the Concept1 device. The study aims to determine whether the novel formulation has a similar clinical profile as the established formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with asthma
* Aged 18 or above
* Patients using inhaled corticosteroid (with or without long acting beta agonist)
* Patients who demonstrate an increase in FEV1 after inhaling a short acting beta agonist

Exclusion Criteria:

* Asthma exacerbations in previous 6 months
* COPD or other pulmonary disease
* Excessive use of short acting beta agonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Wiesbaden, Germany, Germany
- Novartis Investigative Site, Machester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment Period 1: 75 µg indacaterol maleate (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 2: placebo to indacterol (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 3: placebo to indacaterol (lactose blend) + 75 µg indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 4: placebo to indacaterol (lactose blend) + 37.5 µg Indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. All participants took part in a 7 day run-in period. There was a minimum 14 day washout between each treatment period. Participants continued their current treatment with Inhaled corticosteroids. Inhaled short-acting B2-agonist salbutamol was available for use as rescue medication throughout the study.
- Sequence 2: Treatment Period 1: placebo to indacaterol (lactose blend) + 75 µg indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 2: 75 µg indacaterol maleate (lactose blend) + placebo to indacterol (PulmoSphereTM ) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 3: placebo to indacaterol (lactose blend) + 37.5 µg Indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 4: placebo to indacterol (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. All participants took part in a 7 day run-in period. There was a minimum 14 day washout between each treatment period. Participants continued their current treatment with Inhaled corticosteroids. Inhaled short-acting B2-agonist salbutamol was available for use as rescue medication throughout the study.
- Sequence 3: Treatment Period 1: placebo to indacaterol (lactose blend) + 37.5 µg Indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 2: placebo to indacaterol (lactose blend) + 75 µg indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 3: placebo to indacterol (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 4: 75 µg indacaterol maleate (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. All participants took part in a 7 day run-in period. There was a minimum 14 day washout between each treatment period. Participants continued their current treatment with Inhaled corticosteroids. Inhaled short-acting B2-agonist salbutamol was available for use as rescue medication throughout the study.
- Sequence 4: Treatment Period 1: placebo to indacterol (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 2: placebo to indacaterol (lactose blend) + 37.5 µg Indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 3: 75 µg indacaterol maleate (lactose blend) + placebo to indacterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. Treatment Period 4: placebo to indacaterol (lactose blend) + 75 µg indacaterol (PulmoSphereTM) delivered via the Concept1 device once daily in the morning for 7 days. All participants took part in a 7 day run-in period. There was a minimum 14 day washout between each treatment period. Participants continued their current treatment with Inhaled corticosteroids. Inhaled short-acting B2-agonist salbutamol was available for use as rescue medication throughout the study.
Period: Treatment Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 9 | 9 | 9
Completed | 8 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 (1 patient completed Period 1 but did not enter Period 2 due to a Protocol deviation.) | 8 (1 patient completed Period 1 but did not enter Period 2 due to an Adverse event (AE).) | 9 | 9
Completed | 7 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Subject withdrew consent | 0 | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 8 | 9 | 8
Completed | 7 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 8 | 9 | 6 (2 patients completed Period 3 but did not enter Period 4 due to a Protocol deviation and an AE.)
Completed | 7 | 8 | 9 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to one of four treatment sequences.
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) After 7 Days of Treatment
Description: Spirometry was performed according to internationally accepted standards at Day 8. Trough FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Trough FEV1 was defined as the average of the FEV1 measurements at 23 hours 10 minutes and 23 hours 45 minutes post dose.at Day 8. Analysis of Covariance with treatment, period, sequence and subject nested within sequence as fixed effects and period FEV1 baseline as a covariate.
Time Frame: Day 8
Population: Pharmacodynamics Analysis set included all participants that received at least one dose of study drug and had baseline and at least one post-baseline FEV1 measurement.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- 75 µg Indacaterol (LB): 75 µg indacaterol lactose blend (LB) delivered via the Concept1 device once daily in the morning for 7 days.
- 75 µg Indacaterol (PoS): 75 µg indacaterol PulmoSphereTM (PoS) delivered via the Concept1 device daily in the morning for 7 days.
- 37.5 µg Indacaterol (PoS): 37.5 µg indacaterol PulmoSphereTM (PoS) delivered via the Concept1 device in the morning for 7 days.
- Placebo: Placebo to indacterol lactose blend or PulmoSphereTM delivered via the Concept1 device in the morning for 7 days.
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 33 | 30 | 32 | 33
Liters | 2.84 (0.03) | 2.83 (0.03) | 2.80 (0.03) | 2.64 (0.03)

2. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) After 1 Day of Treatment
Description: Spirometry was performed according to internationally accepted standards at Day 2. Trough FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Trough FEV1 was defined as the average of the FEV1 measurements at 23 hours 10 minutes and 23 hours 45 minutes post dose at Day 2. Analysis of Covariance with treatment, period, sequence and subject nested within sequence as fixed effects and period FEV1 baseline as a covariate.
Time Frame: Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Liters | 2.83 (0.03) | 2.84 (0.03) | 2.81 (0.03) | 2.62 (0.03)

3. Secondary Outcome: Peak FEV1 at Day 1 and Day 7
Description: Spirometry was performed according to internationally accepted standards at 0, 15 and 30 minutes; 1,2,3,4,8,12 hours on Day 1 and 23.16 and 23.75 hours on Day 2 after 1 day of treatment and on Day 7 and Day 8 following 7 days of treatment. Peak FEV1 was the maximum FEV1 post treatment. Analysis of Covariance with treatment, period, sequence and subject nested within sequence as fixed effects and period FEV1 baseline included as a covariate.
Time Frame: Day 1, Day 7
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Liters
  Day 1 | 3.08 [3.04 to 3.13] | 3.11 [3.07 to 3.16] | 3.05 [3.01 to 3.10] | 2.85 [2.80 to 2.89]
  Day 7 (n=33,30,32,33) | 3.09 [3.05 to 3.13] | 3.11 [3.06 to 3.15] | 3.10 [3.06 to 3.14] | 2.89 [2.85 to 2.93]

4. Secondary Outcome: Time to Peak FEV1 at Day 1 and Day 7
Description: Spirometry was performed according to internationally accepted standards. Time to the peak (maximum) FEV1 is recorded. Analysis of Covariance with treatment, period, sequence and subject nested within sequence as fixed effects and period FEV1 baseline as a covariate.
Time Frame: Day 1, Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Hours
  Day 1 | 3.98 [0.25 to 23.77] | 3.02 [0.25 to 23.75] | 3.00 [0.25 to 23.75] | 3.00 [0.25 to 24.77]
  Day 7 (n=33,30,32,33) | 3.00 [0.22 to 23.82] | 3.05 [0.25 to 23.77] | 3.00 [0.98 to 23.78] | 3.97 [0.25 to 23.77]

5. Secondary Outcome: FEV1 at Each Time-Point on Day 1 and Day 2
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8, 12 hours on Day 1 and 23.16 and 23.75 hours on Day 2. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Day 1, Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Liters
  0 minutes post-dose | 2.61 (0.71) | 2.65 (0.70) | 2.68 (0.68) | 2.67 (0.69)
  5 minutes post-dose | 2.85 (0.76) | 2.97 (0.80) | 2.90 (0.75) | 2.66 (0.69)
  30 minutes post-dose | 2.86 (0.76) | 2.96 (0.75) | 2.93 (0.73) | 2.70 (0.71)
  1 hour post-dose | 2.89 (0.76) | 3.03 (0.80) | 2.95 (0.75) | 2.73 (0.72)
  2 hours post-dose | 2.98 (0.73) | 3.06 (0.81) | 3.02 (0.74) | 2.82 (0.68)
  3 hours post-dose | 2.98 (0.76) | 3.09 (0.80) | 3.05 (0.75) | 2.80 (0.69)
  4 hours post-dose | 2.99 (0.73) | 3.07 (0.81) | 3.00 (0.75) | 2.77 (0.67)
  8 hours post-dose | 2.80 (0.60) | 2.99 (0.83) | 2.89 (0.79) | 2.70 (0.68)
  12 hours post-dose | 2.74 (0.65) | 2.92 (0.79) | 2.85 (0.79) | 2.71 (0.67)
  23.16 hours post-dose | 2.81 (0.74) | 2.85 (0.77) | 2.83 (0.76) | 2.59 (0.69)
  23.75 hours post-dose | 2.89 (0.75) | 2.88 (0.80) | 2.85 (0.72) | 2.68 (0.69)

6. Secondary Outcome: FEV1 at Each Time-Point on Day 7 and Day 8
Description: Spirometry was conducted according to internationally accepted standards at 0, 15 and 30 minutes; 1,2,3,4,8,12 hours on Day 7 and 23.16 and 23.75 hours on Day 8. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Day 7, Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 33 | 30 | 32 | 33
Liters
  0 minutes post-dose | 2.80 (0.77) | 2.79 (0.72) | 2.85 (0.73) | 2.63 (0.67)
  15 minutes post-dose | 2.87 (0.80) | 2.88 (0.77) | 2.92 (0.76) | 2.65 (0.72)
  30 minutes post-dose | 2.91 (0.79) | 2.92 (0.76) | 2.94 (0.77) | 2.64 (0.72)
  1 hour post-dose | 2.94 (0.75) | 2.96 (0.77) | 2.97 (0.76) | 2.72 (0.70)
  2 hours post-dose | 2.99 (0.76) | 3.00 (0.72) | 3.00 (0.73) | 2.79 (0.72)
  3 hours post-dose | 2.99 (0.74) | 2.99 (0.75) | 3.06 (0.75) | 2.79 (0.72)
  4 hours post-dose | 2.98 (0.75) | 2.98 (0.73) | 3.02 (0.70) | 2.78 (0.70)
  8 hours post-dose | 2.82 (0.64) | 2.88 (0.77) | 2.89 (0.75) | 2.76 (0.65)
  12 hours post-dose | 2.76 (0.66) | 2.80 (0.78) | 2.82 (0.76) | 2.65 (0.70)
  23.16 hours post-dose | 2.79 (0.71) | 2.79 (0.77) | 2.79 (0.79) | 2.64 (0.68)
  23.75 hours post-dose | 2.89 (0.72) | 2.87 (0.76) | 2.87 (0.74) | 2.74 (0.68)

7. Secondary Outcome: Forced Vital Capacity (FVC) at Each Time-Point on Day 1 and Day 2
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8 and 12 hours on Day 1 and 23.16 and 23.75 hours on Day 2. FVC is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Day 1, Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Liters
  0 minutes post-dose | 4.11 (1.02) | 4.30 (0.98) | 4.23 (1.03) | 4.27 (1.02)
  15 minutes post-dose | 4.29 (1.07) | 4.52 (1.10) | 4.34 (1.04) | 4.25 (1.03)
  30 minutes post-dose | 4.29 (1.03) | 4.47 (1.02) | 4.39 (1.01) | 4.18 (1.07)
  1 hour post-dose | 4.33 (1.06) | 4.49 (1.05) | 4.38 (1.06) | 4.30 (1.06)
  2 hours post-dose | 4.39 (0.99) | 4.54 (1.07) | 4.45 (1.02) | 4.36 (0.97)
  3 hours post-dose | 4.38 (1.04) | 4.52 (1.05) | 4.44 (0.98) | 4.33 (0.98)
  4 hours post-dose | 4.39 (1.01) | 4.54 (1.06) | 4.40 (1.01) | 4.30 (0.98)
  8 hours post-dose | 4.20 (0.86) | 4.51 (1.09) | 4.35 (1.07) | 4.21 (1.01)
  12 hours post-dose | 4.16 (0.93) | 4.42 (1.05) | 4.29 (1.04) | 4.24 (1.02)
  23.16 hours post-dose | 4.34 (1.06) | 4.44 (1.08) | 4.31 (1.08) | 4.21 (0.99)
  23.75 hours post-dose | 4.41 (1.06) | 4.41 (1.10) | 4.36 (1.08) | 4.30 (0.99)

8. Secondary Outcome: Forced Vital Capacity (FVC) at Each Time-Point on Day 7 and Day 8
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8 and 12 hours on Day 7 and 23.16 and 23.75 hours on Day 8. FVC is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Day 7, Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 33 | 30 | 32 | 33
Liters
  0 minutes post-dose | 4.28 (1.07) | 4.30 (0.93) | 4.35 (1.06) | 4.22 (1.00)
  15 minutes post-dose | 4.34 (1.09) | 4.33 (0.95) | 4.36 (1.06) | 4.21 (1.04)
  30 minutes post-dose | 4.36 (1.08) | 4.36 (0.96) | 4.37 (1.06) | 4.21 (1.04)
  1 hour post-dose | 4.37 (1.06) | 4.35 (0.97) | 4.41 (1.05) | 4.28 (1.03)
  2 hours post-dose | 4.39 (1.04) | 4.40 (0.90) | 4.42 (1.02) | 4.37 (1.06)
  3 hours post-dose | 4.37 (1.01) | 4.40 (0.93) | 4.46 (1.03) | 4.34 (1.05)
  4 hours post-dose | 4.38 (1.05) | 4.39 (0.91) | 4.44 (0.99) | 4.32 (1.03)
  8 hours post-dose | 4.24 (0.97) | 4.29 (0.94) | 4.31 (1.05) | 4.31 (1.01)
  12 hours post-dose | 4.17 (0.98) | 4.23 (0.94) | 4.25 (1.04) | 4.21 (1.03)
  23.16 hours post-dose | 4.32 (1.08) | 4.30 (0.97) | 4.29 (1.08) | 4.28 (1.02)
  23.75 hours post-dose | 4.41 (1.08) | 4.34 (0.97) | 4.34 (1.08) | 4.36 (1.02)

9. Secondary Outcome: FEV1/FVC at Each Post-Dose Time Point on Day 1 and Day 2
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8 and 12 hours on Day 1 and 23.16 and 23.75 hours on Day 2. FEV1/FVC ratio is the percentage of the total FVC that is expelled from the lungs during the first second of forced exhalation.
Time Frame: Day1, Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 34 | 34 | 34
Ratio
  0 minutes post-dose | 0.63 (0.08) | 0.62 (0.08) | 0.64 (0.09) | 0.63 (0.09)
  15 minutes post-dose | 0.67 (0.08) | 0.66 (0.07) | 0.67 (0.09) | 0.63 (0.09)
  30 minutes post-dose | 0.67 (0.07) | 0.66 (0.07) | 0.67 (0.08) | 0.65 (0.09)
  1 hour post-dose | 0.67 (0.07) | 0.67 (0.07) | 0.68 (0.08) | 0.64 (0.08)
  2 hours post-dose | 0.68 (0.08) | 0.67 (0.07) | 0.68 (0.08) | 0.65 (0.08)
  3 hours post-dose | 0.68 (0.08) | 0.68 (0.07) | 0.69 (0.08) | 0.65 (0.08)
  4 hours post-dose | 0.68 (0.08) | 0.67 (0.07) | 0.68 (0.08) | 0.65 (0.08)
  8 hours post-dose | 0.67 (0.07) | 0.66 (0.07) | 0.67 (0.08) | 0.64 (0.07)
  12 hours post-dose | 0.66 (0.08) | 0.66 (0.07) | 0.66 (0.08) | 0.64 (0.08)
  23.16 hours post-dose | 0.65 (0.09) | 0.64 (0.08) | 0.66 (0.09) | 0.62 (0.09)
  23.75 hours post-dose | 0.66 (0.08) | 0.65 (0.08) | 0.66 (0.08) | 0.63 (0.08)

10. Secondary Outcome: FEV1/FVC at Each Post-dose Time Point on Day 7 and Day 8
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8 and 12 hours on Day 1 and 23.16 and 23.75 hours on Day 2 after treatment. FEV1/FVC ratio is the percentage of the total FVC that is expelled from the lungs during the first second of forced exhalation.
Time Frame: Day 7, Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 33 | 30 | 32 | 33
Ratio
  0 minutes post-dose | 0.65 (0.08) | 0.65 (0.07) | 0.65 (0.08) | 0.62 (0.08)
  15 minutes post-dose | 0.66 (0.08) | 0.66 (0.07) | 0.67 (0.07) | 0.63 (0.08)
  30 minutes post-dose | 0.67 (0.08) | 0.67 (0.06) | 0.67 (0.07) | 0.63 (0.09)
  1 hour post-dose | 0.67 (0.07) | 0.68 (0.07) | 0.67 (0.07) | 0.64 (0.08)
  2 hours post-dose | 0.68 (0.07) | 0.68 (0.06) | 0.68 (0.07) | 0.64 (0.08)
  3 hours post-dose | 0.68 (0.07) | 0.68 (0.07) | 0.69 (0.08) | 0.65 (0.09)
  4 hours post-dose | 0.68 (0.07) | 0.68 (0.07) | 0.68 (0.07) | 0.64 (0.08)
  8 hours post-dose | 0.66 (0.07) | 0.67 (0.07) | 0.67 (0.08) | 0.64 (0.08)
  12 hours post-dose | 0.66 (0.08) | 0.66 (0.07) | 0.66 (0.08) | 0.63 (0.08)
  23.16 hours post-dose | 0.64 (0.67) | 0.65 (0.08) | 0.65 (0.08) | 0.62 (0.09)
  23.75 hours post-dose | 0.65 (0.72) | 0.66 (0.07) | 0.66 (0.08) | 0.63 (0.09)

11. Secondary Outcome: Forced Expiratory Flow 25- 75% (FEF25-75) on Day 1 and Day 2
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8 and 12 hours on Day 1 and 23.16 and 23.75 hours on Day 2. The forced expiratory flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry.
Time Frame: Day 1, Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/second
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Liters/second
  0 minutes post-dose | 1.55 (0.68) | 1.52 (0.70) | 1.54 (0.67) | 1.56 (0.71)
  15 minutes post-dose | 1.78 (0.75) | 1.81 (0.79) | 1.82 (0.77) | 1.54 (0.72)
  30 minutes post-dose | 1.80 (0.80) | 1.82 (0.77) | 1.84 (0.73) | 1.61 (0.74)
  1 hour post-dose | 1.79 (0.77) | 1.95 (0.85) | 1.89 (0.75) | 1.59 (0.73)
  2 hours post-dose | 1.90 (0.80) | 1.93 (0.84) | 1.92 (0.79) | 1.68 (0.74)
  3 hours post-dose | 1.89 (0.81) | 2.01 (0.83) | 1.99 (0.85) | 1.68 (0.77)
  4 hours post-dose | 1.94 (0.82) | 1.94 (0.85) | 1.92 (0.80) | 1.65 (0.70)
  8 hours post-dose | 1.71 (0.69) | 1.83 (0.84) | 1.79 (0.81) | 1.59 (0.66)
  12 hours post-dose | 1.63 (0.65) | 1.77 (0.78) | 1.76 (0.83) | 1.61 (0.69)
  23.16 hours post-dose | 1.70 (0.77) | 1.68 (0.75) | 1.78 (0.80) | 1.51 (0.70)
  23.75 hours post-dose | 1.77 (0.74) | 1.76 (0.77) | 1.75 (0.71) | 1.56 (0.71)

12. Secondary Outcome: Forced Expiratory Flow 25- 75% (FEF25-75) on Day 7 and Day 8
Description: Spirometry was conducted according to internationally accepted standards post-dose at 0, 15 and 30 minutes; 1, 2, 3, 4, 8 and 12 hours on Day 7 and 23.16 and 23.75 hours on Day 8. The forced expiratory flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry.
Time Frame: Day 7, Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/second
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 33 | 30 | 32 | 33
Liters/second
  0 minutes post-dose | 1.70 (0.75) | 1.69 (0.76) | 1.71 (0.78) | 1.51 (0.67)
  15 minutes post-dose | 1.76 (0.83) | 1.78 (0.82) | 1.83 (0.80) | 1.54 (0.73)
  30 minutes post-dose | 1.80 (0.79) | 1.80 (0.82) | 1.83 (0.81) | 1.57 (0.72)
  1 hour post-dose | 1.82 (0.77) | 1.89 (0.84) | 1.87 (0.80) | 1.61 (0.69)
  2 hours post-dose | 1.88 (0.80) | 1.89 (0.77) | 1.91 (0.82) | 1.64 (0.72)
  3 hours post-dose | 1.91 (0.80) | 1.88 (0.81) | 2.02 (0.82) | 1.69 (0.70)
  4 hours post-dose | 1.90 (0.82) | 1.88 (0.82) | 1.93 (0.83) | 1.65 (0.73)
  8 hours post-dose | 1.71 (0.66) | 1.80 (0.82) | 1.81 (0.82) | 1.64 (0.67)
  12 hours post-dose | 1.66 (0.68) | 1.68 (0.83) | 1.76 (0.83) | 1.56 (0.72)
  23.16 hours post-dose | 1.66 (0.67) | 1.69 (0.81) | 1.68 (0.84) | 1.52 (0.64)
  23.75 hours post-dose | 1.74 (0.72) | 1.73 (0.79) | 1.79 (0.76) | 1.62 (0.72)

13. Secondary Outcome: Standardized FEV1 AUC Between Baseline (Pre-dose) and 4 Hour Post-dose (AUC0-4h)
Description: Spirometry was conducted according to internationally accepted standards at predose, 5, 15 and 30 minutes, 1, 2 and 4 hours post-dose on Day 1 and Day 7. The standardized (with respect to the length of time) area under the curve (AUC) for FEV1 was calculated using trapezoidal rule between 5 min and 4 h post. Analysis of Covariance with treatment, period, sequence and subject nested within sequence as fixed effects and period FEV1 baseline as a covariate.
Time Frame: Day 1, Day 7
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 30 | 33
Liters
  Day 1 | 2.94 [2.90 to 2.99] | 3.00 [2.95 to 3.05] | 2.94 [2.89 to 2.99] | 2.72 [2.68 to 2.77]
  Day 7 (n=33,30,32,33) | 2.96 [2.92 to 3.00] | 2.98 [2.93 to 3.02] | 2.97 [2.93 to 3.02] | 2.73 [2.68 to 2.77]

14. Secondary Outcome: Standardized FEV1 AUC Between Baseline (Pre-dose) and 12 Hour Post-dose (AUC0-12h)
Description: Spirometry was conducted according to internationally accepted standards at predose, 5 , 15 and 30 min, 1, 2, 4, 8 and 12 hours post-dose on Day 1 and Day 7. The standardized (with respect to the length of time) area under the curve (AUC) for FEV1 was calculated using trapezoidal rule between 5 min and 12 h post. Analysis of covariance with treatment, period, sequence and subject nested within sequence as fixed effects and FEV1 period baseline as a covariate.
Time Frame: Day 1, Day 7
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Liters
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 32 | 29 | 30 | 31
Liters
  Day 1 | 2.90 [2.85 to 2.95] | 2.94 [2.89 to 2.99] | 2.87 [2.82 to 2.92] | 2.68 [2.63 to 2.72]
  Day 7 (n=31,29,30,31) | 2.93 [2.88 to 2.97] | 2.92 [2.88 to 2.96] | 2.91 [2.87 to 2.95] | 2.70 [2.66 to 2.74]

15. Secondary Outcome: Peak Expiratory Flow Rate in the Morning in the Evening
Description: PEFR was measured on all days from Screening Visit 2 to end of study visit: twice daily pre-dose (prior to Inhaled Corticosteroids) and approximately 12 hours post-dose (during the treatment period). Each subject was provided with a PEFR meter and recorded the PEFR readings in a daily diary. repeated measures. Analysis of covariance with treatment, period, sequence, day and treatment-day interaction as fixed effect and subject as a random effect and baseline PEFR as a covariate in the model.
Time Frame: Up to 101 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters per second
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Liters per second
  Morning | 451.33 (2.35) | 447.15 (2.50) | 444.11 (2.47) | 421.58 (2.41)
  Evening | 474.09 (2.18) | 464.39 (2.33) | 463.28 (2.30) | 433.60 (2.24)

16. Secondary Outcome: Number of Puffs of Rescue Medicine
Description: Salbutamol (100 µg/puff) was used as rescued medicine. The total number of puffs per day was calculated and divided by the number of days with data to determine the mean daily number of puffs of rescue medication for each patient and was recorded in the patient diary from Baseline until Day 8 of Treatment Period 4. Analysis of covariance with treatment, period, sequence, and subject nested within sequence as fixed effect.
Time Frame: Up to 101 days
Population: Participants in the Pharmacodynamics Analysis set (included all participants that received at least one dose of study drug and had baseline and at least one post-baseline FEV1 measurement) who used rescue medication.
Measure: Least Squares Mean (90% Confidence Interval); unit: Puffs/day
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 13 | 14 | 8 | 16
Puffs/day | 1.98 [1.90 to 2.06] | 1.90 [1.83 to 1.98] | 1.91 [1.82 to 2.00] | 1.94 [1.87 to 2.00]

17. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Adverse event are defined as any unfavorable and unintended diagnosis, symptoms, sign (including an abnormal lab finding), syndrome or disease which either occurs during the study, having been absent at baseline, or if present at baseline appear to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization , cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgments of the investigators represent significant hazards. Additional information about adverse events can be found in the Adverse Event section
Time Frame: Up to 101 days
Population: Safety population inlcuded all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Number analyzed (Participants) | 34 | 31 | 33 | 33
Participants | 14 | 16 | 17 | 10

18. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) After Drug Administration
Time Frame: Day1, Day 7
Population: PK Analysis Set
Measure: Median (Full Range); unit: Hours
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS)
Number analyzed (Participants) | 34 | 31 | 33
Hours
  Day 1 (n=31,30,31) | 0.27 [0.22 to 1.03] | 0.48 [0.20 to 0.58] | 0.48 [0.20 to 1.00]
  Day 7 (n=33,31,31) | 0.25 [0.08 to 0.75] | 0.48 [0.22 to 0.98] | 0.25 [0.22 to 1.02]

19. Secondary Outcome: Observed Maximum Concentration (Cmax) After Drug Administration
Time Frame: Day 1, Day 7
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS)
Number analyzed (Participants) | 34 | 31 | 33
pg/mL
  Day 1 (n=31,30,31) | 72.9 (25.7) | 124 (55.7) | 64.2 (27.9)
  Day 7 (n=33,31,31) | 112 (27.1) | 174 (61.4) | 90.5 (23.9)

20. Secondary Outcome: Area Under the Curve Pre-dose to 24 Hour Post Dose (AUC0-24h)
Time Frame: Day 1, Day 7
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: hour*pg/mL
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS)
Number analyzed (Participants) | 34 | 31 | 33
hour*pg/mL
  Day 1 (n=30,30,27) | 501 (149) | 802 (308) | 451 (134)
  Day 7 (n=33,31,31) | 1110 (273) | 1770 (522) | 952 (287)

ADVERSE EVENTS:
Description: The number of participants at risk for serious adverse events and non-serious adverse events is based on those participants in the arm who received at least one dose of study drug.
Arm/Group | 75 µg Indacaterol (LB) | 75 µg Indacaterol (PoS) | 37.5 µg Indacaterol (PoS) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 14/34 | 16/31 | 17/33 | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 75 µg Indacaterol (LB) (N=34) | 75 µg Indacaterol (PoS) (N=31) | 37.5 µg Indacaterol (PoS) (N=33) | Placebo (N=33)
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 75 µg Indacaterol (LB) (N=34) | 75 µg Indacaterol (PoS) (N=31) | 37.5 µg Indacaterol (PoS) (N=33) | Placebo (N=33)
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Product taste abnormal (General disorders) | 0 | 0 | 2 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 4 | 5 | 5
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 8 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.